CLINICAL TRIAL: NCT05052177
Title: Percutaneous Edge To Edge Repair for the Treatment of Severe Tricuspid Valve Regurgitation in High-surgical Risk Patients With Systemic Right Ventricle : a Multicentric French Cohort.
Brief Title: Percutaneous Edge To Edge Repair for the Treatment of Severe Tricuspid Valve Regurgitation in High-surgical Risk Patients With Systemic Right Ventricle : a Multicentric French Cohort (PETER-TRESRIV)
Acronym: PETER-TRESRIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Alexandre Silini, Intern, University of Bordeaux
Other Study IDs: University of Bordeaux
Record Dates: First submitted 2021-09-02; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Systemic Right Ventricle; Tricuspid Regurgitation; Congenital Heart Disease
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patient with systemic right ventricles with severe tricuspid regurgitation and high surgical risk: * inclusion criteria:
    * > 18-years-old
    * Right systemic ventricle
    * Severe tricuspid regurgitation
    * Symptomatic patient (NYHA 2 - 4) despite optimal medical therapy
    * High-risk surgical patient deemed not eligible for surgery by a multi-disciplinary and thus having underwent a percutaneous treatment of tricuspid regurgitation
  * exclusion criteria - pregnant ou breastfeeding women
  Interventions: Device: Edge to edge repair in systemic tricuspid valve regurgitation

INTERVENTIONS:
Device: Edge to edge repair in systemic tricuspid valve regurgitation — Edge to edge repair of severe tricuspid regurgitation on a right systemic ventricle with a Mitraclip device.

SUMMARY:
Our study is about to follow adult congenital patients, known with systemic right ventricle (mostly correct transposition of the great arteries ou congenitally corrected transposition fo the great arteries) and systemic valve severe regurgitation which was treated with a Mitraclip device on this tricuspid valve.

It's an observationnal study with a 2 years follow up with clinical (symptoms, complications, VO2 exercice test) echographic and MRI outcomes

.

DETAILED DESCRIPTION:
Patients with systemic right ventricle (mostly congenitally-corrected transposition of the great arteries or transposition of the great arteries corrected by atrial switch) commonly develop significant systemic tricuspid valve regurgitation which is a therapeutic dilemma for the care team. Surgery (valvuloplasty or replacement) is the common and historical treatment but the rate of mortality is high and results about long-term benefit are contradicting. Percutaneous edge to edge repair could be a alternative to surgery.

10 high-risk surgical patients with severe systemic tricuspid regurgitation undergoing a percutaneous repair were included between January 2019 and November 2022. Our study is a retrospective analysis of short and mid-term clinical, biological, echocardiographic and MRI/TDM outcomes with an expected minimum follow-up of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* > 18-years-old
* Right systemic ventricle
* Severe tricuspid regurgitation
* Symptomatic patient (NYHA 2 - 4) despite optimal medical therapy
* High-risk surgical patient deemed not eligible for surgery by a multi-disciplinary and thus having underwent a percutaneous treatment of tricuspid regurgitation

Exclusion Criteria:

* pregnant
* breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic right ventricle who underwent a percutaneous edge to edge systemic valve repair for the treatment of severe tricuspid valve regurgitation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical, VO2 max testing, biological, echocardiographic, cross-sectionnal Imaging data. | 2 years
  Clinical data : dyspnea (NYHA 1/2/3/4), heart palpitations (yes/no), heart failure in the 6 previous months (yes/no)
VO2 max testing data. | 2 years
  VO2 max testing: VO2 max (ml/min/kg), strenght in watts
Biological data. | 2 years
  Biological data : hemoglobine (g/dL), hematocrit (%), creatinine (µmol/L), BNP/nt-proBNP (ng/mL) at baseline, 6, 12, 24 months
Echographic data. | 2 years
  Echocardiographic data : tricuspid insuffisency severity (régurgitant orifice area in mm²), régurgitant volume (mL)), tricuspid annular diameter (cm), and right ventricle systemic function (S'VD in cm/s, TAPSE in mm, shortening right ventricle fraction in %), and area (end-diastolic and end-systolic area) at baseline, 6, 12, 24 months
Cross-sectionnal Imaging data. | 2 years
  Cross-sectionnal imaging data : quantitative parameters of tricuspid regurgitation (regurgitant volume in mL, percentage of regurgitation in %) and right ventricle systemic function (ejection fraction in %) and volume (end-diastolic and end-systolic volume in mL) at baseline and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre SILINI, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Filippov AA, del Nido PJ, Vasilyev NV. Management of Systemic Right Ventricular Failure in Patients With Congenitally Corrected Transposition of the Great Arteries. Circulation. 25 oct 2016;134(17):1293-302. — https://pubmed.ncbi.nlm.nih.gov/27777298/